CLINICAL TRIAL: NCT04645121
Title: Carbon Monoxide-based Rebreathing Method and Bioimpedance to Assess Intra- and Extravascular Volume in Hemodialysis Patients
Brief Title: Carbon Monoxide-based Rebreathing Method and Bioimpedance in Hemodialysis Patients
Acronym: HEMOVOL
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Bo Feldt-Rasmussen, Professor, Rigshospitalet, Denmark
Other Study IDs: H-20031445
Record Dates: First submitted 2020-11-22; First posted 2020-11-27 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Hemodialysis Complication; Volume Overload
MeSH Terms: conditions — Edema | interventions — Albumins

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemodialysis group: Subjects receiving maintenance hemodialysis for at least three months
  Interventions: Device: Carbon Monoxide-based Rebreathing; Device: Bioimpedance; Radiation: Radioactive labelling of erythrocytes and albumin
- Case group: Healthy subjects with eGFR above 60 ml/min/1.73m2
  Interventions: Device: Carbon Monoxide-based Rebreathing; Device: Bioimpedance; Radiation: Radioactive labelling of erythrocytes and albumin

INTERVENTIONS:
Device: Carbon Monoxide-based Rebreathing — 6 minutes Carbon Monoxide-based Rebreathing that estimate blood volume, plasma volume and erythrocyte volume.
Device: Bioimpedance — Measures total volume, intra and extracellular volume.
Radiation: Radioactive labelling of erythrocytes and albumin — Measure blood volume, plasma volume and erythrocyte volume.

SUMMARY:
The study is a case-control study with the primary aim of objectifying the volume status of patients receiving hemodialysis. Volume status will be assessed at dry weight and evaluated by a carbon monoxide rebreathing method, that measures blood volume, and bioimpedance that measures total body water. Case-control subjects will be matched on gender, age and weight.

Secondary aims are to evaluate the carbon monoxide rebreathing method. Blood volumes obtained by the carbon monoxide rebreathing method will be correlated to blood volumes obtained by radioactive labelling of erythrocytes and albumin. In addition, it will be investigated whether hemoglobin is a valid marker of anemia in patients receiving hemodialysis by measuring the erythrocyte volume and the hemoglobin mass by the carbon monoxide rebreathing method and correlating this to the hemoglobin concentration measured before and after dialysis.

DETAILED DESCRIPTION:
Aim:

1. To combine a carbon monoxide rebreathing method and bioimpedance which allows to objectively measure the amount of fluid in the bloodstream (intravascular) and throughout the body, and thereby test the actual amount of fluid in the body when patients are hydrated according to their clinical dry weight.
2. To validate carbon monoxide rebreathing method in hemodialysis patients compared against a radioactive labeling of erythrocytes and albumin (the gold standard).
3. To investigate whether hemoglobin is a valid marker of anemia in this patient population by measuring the erythrocyte volume and hemoglobin mass by the carbon monoxide rebreathing method and correlating this to the hemoglobin concentration.

Background:

Anemia and overhydration are challenging conditions in patients on hemodialysis. Overhydration is associated with hypertension, cardiomyopathy and increased mortality. In assessing the patient's volume status, blood pressure, body weight and peripheral edema are used as indicators. To achieve a more accurate estimate, these measures have been combined with various techniques, such as relative changes in blood volume (measured with blood volume sensor (BVS)) and bioimpedance. These methods are used to varying degrees in everyday clinical practice.

In case of overhydration, fluid is distributed intravascularly and can thereby expand blood volume. The primary clinical problem with an expanded blood volume is hypertension and increased risk of cardiovascular complications. Measurement of the intravascular volume can therefore have great clinical relevance, but currently there are no direct measures for this implemented in the clinical daily routine. Various techniques have been used for research purposes. These include fluorescent dilution techniques, radioactive labeling of erythrocytes and albumin, as well as infusion of dialysate during dialysis where changes in BVS measurements can be used to calculate the intravascular volumes.

Bioimpedance can be used to measure the total water phase and the intra- and extracellular volume. The method has been shown to be useful in the diagnosis of overhydration in hemodialysis patients. Overhydration detected by bioimpedance in hemodialysis patients has been shown to correlate to increased mortality. Bioimpedance is a non-invasive, painless and practically useful way of assessing the volume status.

Anemia is another significant challenge in patients on hemodialysis. The majority of patients on hemodialysis have a significant decrease in endogenous erythropoietin production, which causes anemia and requires treatment with an erythrocyte stimulant (ESA). The basis for anemia diagnosis and the decision on ESA treatment in hemodialysis patients is based on pre-dialysis hemoglobin (measured at dialysis start-up). Upon overhydration, fluid distributed to the intravascular space will lead to dilated plasma volume (PV) and dilution of hemoglobin. This dilution and thus artificial decrease in hemoglobin makes pre-dialysis hemoglobin difficult to interpret in patients on dialysis. Time-averaged hemoglobin, calculated on the basis of pre-dialysis and post-dialysis hemoglobin, has been shown to correlate better with the actual hemoglobin of hemodialysis patients, but the value has not gained ground in practice.

The carbon monoxide rebreathing method is a well-proven technique for determining intravascular volume, (blood volume, BV), PV and red blood cell volume (RBCV). In renally healthy patients, the method is validated against a radioactive labeling technique (gold standard) where high correlation (r = 0.97) has been demonstrated between the two methods. The carbon monoxide rebreathing method has also been shown to be able to detect even very small changes in blood volume. The method is safe and requires 6 minutes of carbon monoxide inhalation. A prerequisite for using the carbon monoxide rebreathing method is a normal diffusion of gas over the lungs, which allows uptake into the blood. Dialysis patients may be significantly overhydrated and possible accumulation of water in the alveoli may decrease the diffusion of carbon monoxide and affect the method. Against this background, the method is to be validated against a radioactive labeling technique.

The validity of the carbon monoxide rebreathing method in hemodialysis patients has not been performed which is important if the method is to be implemented clinically and for research purposes.

Method:

Case-control study with 25 patients in each group. The case group consists of hemodialysis patients and the control group consists of healthy individuals with eGFR above 60 ml/min/1.73m2. Subjects were matched on gender, age (+/- 5 years) and (weight +/- 10kg).

Hemodialysis group: 25 hemodialysis patients are included. Immediately before the start of dialysis, the total body water is measured by bioimpedance and blood samples are taken. A normal hemodialysis lasts 3-4 hours and during this period the patient undergoes fluid extraction corresponding to their estimated dry weight. 30 minutes after the dialysis is completed, the total boby water is measured with bioimpedance and the blood volume, plasma volume and erythrocyte volume are measured by carbon monoxide rebreathing method. In 10 participants, blood volume, plasma volume and the erythrocyte volume are measured by a radioactive labeling of erythrocytes and albumin, where blood is taken at the beginning of dialysis and cleaned at the end of dialysis. Hemoglobin and hematocrit are measured pre-dialysis, post-dialysis and 30 minutes after cessation of dialysis. Participation in the study involving the radioactive labeling of erythrocytes and albumin may be omitted if a participant does not wish the study.

Control group: Includes 25 patients with eGFR above 60 ml/min/1.73m2 and without severe heart failure, liver failure or lung disease. In all participants, the intravascular volume is measured by carbon monoxide rebreathing method and the total body water by bioimpedance. In 10 participants, blood volume is measured by a radioactive label of erythrocytes and albumin. Hemoglobin and other standard samples are measured.

If a participant after inclusion must be withdrawn, the patient is replaced by a new participant until a number of 25 participants in each group is achieved. If a matched participant cannot be found for an included participant, the person in question is withdrawn and replaced by a new one.

Statistics:

Blood volume in patients hemodialysis has been found to be 73.4 ml / kg (SD 15 ml / kg) and from the predicted normal blood volume has been found to be 59.0 ml / kg (SD 9.3 ml / kg). In a two-sided unpaired t-test with α = 0.05, SD = 15 and a power of 90%, a sample size of 23 patients in each group will show a significant difference. A dropout rate of approximately 2 patients is assumed and a total of 25 are included in each group.

After completion of the study and data completion the results are analysed according to primary and secondary endpoints. Results are reported as mean values with confidence interval or median and interquartile range. Data are analysed with parametric (normally distributed data) or non-parametric statistics (non-normal distributed data). A 95 % confidence interval is accepted as statistically significant (p < 0.05). Analysis are performed as a per protocol analysis.

ELIGIBILITY:
Inclusion criteria for hemodialysis group:

* Man/woman aged 18-90 years
* Hemodialysis treatment for a minimum of 3 months
* BMI 18.5-50 kg/m2

Inclusion criteria for control group:

* Man / woman aged 18-90 years
* Renal function with eGFR above 60ml / min and urine albumin-creatinine ratio below 300mg/g
* BMI: 18.5-50 kg / m2 Control group:

Exclusion criteria for hemodialysis:

* Pregnant or breastfeeding
* Hybrid dialysis (both hemodialysis and peritoneal dialysis simultaneously)
* Chronic obstructive pulmonary disease, asthma or interstitial pulmonary fibrosis
* Pulmonary embolism within 6 months
* Lung cancer or previous lung surgery.

Exclusion criteria for control group:

* Pregnant or breastfeeding
* Known heart failure with Left ventricular ejection fraction ˂ 45%
* Liver failure (Child Pugh Score A, B or C)
* Chronic obstructive pulmonary disease, asthma or interstitial pulmonary fibrosis - Pulmonary embolism within 6 months
* Lung cancer or previous lung surgery. Active cancer
* HbA1c over 60mmol / mol
* Edema (except mild lower leg edema)

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Total number of participants: 50 divided in two Groups:
  * 25 subjects receiving hemodialysis
  * 25 subjects with eGFR above 60 ml/min/1.73m2
  The patients are recruited from the department of Nephrology at Rigshospitalet and Herlev Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Blood volume by carbon monoxide rebreathing method | Day 1
  Blood volume measured by carbon monoxide rebreathing method in ml/kg

SECONDARY OUTCOMES:
Erythrocyte volume by carbon monoxide rebreathing method | Day 1
  Erythrocyte volume measured by carbon monoxide rebreathing method in ml/kg
Plasma volume by carbon monoxide rebreathing method | Day 1
  Plasma volume measured by carbon monoxide rebreathing method in ml/kg
Blood volume by Nadler's formula | Day 1
  Blood volume calculated by Nadler's formula in ml/kg
Erythrocyte volume by Nadler's formula | Day 1
  Erythrocyte volume calculated by Nadler's formula in ml/kg
Plasma volume by Nadler's formula | Day 1
  Plasma volume calculated by Nadler's formula in ml/kg
Blood volume by radioactive labelling of erythrocytes and albumin | Day 1
  Blood volume measured by radioactive labelling of erythrocytes and albumin
Erythrocyte volume by radioactive labelling of erythrocytes | Day 1
  Erythrocyte volume measured by radioactive labelling of albumin
Plasma volume by radioactive labelling of albumin | Day 1
  Plasma volume measured by radioactive labelling of albumin
Hemoglobin mass | Day 1
  Hemoglobin mass measured by carbon monoxide rebreathing method in ml/kg
time-averaged hemoglobin | Day 1
  time-averaged hemoglobin calculated from pre- and post-dialysis hemoglobin
Hemoglobin | Day 1
  measured for the control group
Hemoglobin pre-dialysis | Day 1
  For the hemodialysis the hemoglobin concentration obtained pre-hemodialysis (0-30 min before start)
Hemoglobin pre-dialysis | Day 1
  For the hemodialysis the hemoglobin concentration obtained pre-hemodialysis (0-5 min after hemodialysis)
Hemoglobin rebound after dialysis | Day 1
  For the hemodialysis the hemoglobin concentration obtained post- hemodialysis (30 min after dialysis)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Herlev Hospital, Copenhagen
  - Rigshospitalet, Department of Nephrology, København Ø